CLINICAL TRIAL: NCT02829060
Title: The Endourology Disease Group for Excellence (EDGE) Consortium: A Randomized Trial of Preoperative Prophylactic Antibiotics Prior to Percutaneous Nephrolithotomy in Patients With Moderate Risk of Postoperative Infection
Brief Title: Endourology Disease Group Excellence (EDGE) Consortium: Antibiotics (Abx) for Percutaneous Nephrolithotomy (PCNL) Part 2
Acronym: PNLABXPART2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Roger L Sur, M.D., Professor of Surgery, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 160158
Record Dates: First submitted 2016-05-31; First posted 2016-07-12 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Nephrolithiasis; Urinary Tract Infection (UTI); Sepsis
Keywords: nephrolithiasis; percutaneous nephrolithiasis; urinary tract infection (UTI); Sepsis
MeSH Terms: conditions — Nephrolithiasis; Urinary Tract Infections; Sepsis | interventions — Nitrofurantoin; Gentamicins; Ampicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1a: Indwelling drains (48 hr) (Active Comparator): This group has indwelling urinary tubes/drains and a negative urine culture
  * Nitrofurantoin (Macrobid) 100 mg oral bid for 48 hours prior to surgery
  * All patient receive ampicillin IV (2 g) and gentamicin IV (5 mg/kg) within 120 minutes of surgery start time.
  Interventions: Drug: Gentamicin, 5mg/kg; Drug: Ampicillin 2g; Drug: Nitrofurantoin 100 mg, 48 hrs
- 1b: Indwelling drains (7d) (Active Comparator): This group has indwelling urinary tubes/drains and a negative urine culture
  * Nitrofurantoin (Macrobid) 100 mg oral bid for 7 days prior to surgery
  * All patient receive ampicillin IV (2 g) and gentamicin IV (5 mg/kg) within 120 minutes of surgery start time.
  Interventions: Drug: Nitrofurantoin 100 MG, 7d; Drug: Gentamicin, 5mg/kg; Drug: Ampicillin 2g
- 2a: +UCx with Oral Options (48hr) (Active Comparator): This group has a positive pre-operative urine culture with oral antibiotic options
  * Nitrofurantoin (Macrobid) 100 mg oral bid for 48 hours prior to surgery
  * If patient has previous allergies to Macrobid and/or sensitivity profile indicates Macrobid resistance, then one antibiotic will be provided in the following order: nitrofurantoin > sulfamethoxazole-trimethoprim > doxycycline> ciprofloxacin > cephalexin > cefpodoxime.
  * All patient receive ampicillin IV (2 g) and gentamicin IV (5 mg/kg) within 120 minutes of surgery start time.
  Interventions: Drug: Gentamicin, 5mg/kg; Drug: Ampicillin 2g; Drug: Nitrofurantoin 100 mg, 48 hrs
- 2b: +UCx with Oral Options (7d) (Active Comparator): This group has a positive pre-operative urine culture with oral antibiotic options
  * Nitrofurantoin (Macrobid) 100 mg oral bid for 7 days prior to surgery
  * If patient has previous allergies to Macrobid and/or sensitivity profile indicates Macrobid resistance, then one antibiotic will be provided in the following order: nitrofurantoin > sulfamethoxazole-trimethoprim > doxycycline> ciprofloxacin > cephalexin > cefpodoxime.
  * All patient receive ampicillin IV (2 g) and gentamicin IV (5 mg/kg) within 120 minutes of surgery start time.
  Interventions: Drug: Nitrofurantoin 100 MG, 7d; Drug: Gentamicin, 5mg/kg; Drug: Ampicillin 2g
- 3a: +UCx No Oral options (48hr) (Active Comparator): This group has a positive pre-operative urine culture with no oral antibiotic options based on culture sensitivities
  * 48 hour course of an IV/Intramuscular (IM) antibiotic (proven effective on sensitivity profile)
  * Gentamicin (80 mg) preferred if sensitive
  * All patient receive ampicillin IV (2 g) and gentamicin IV (5 mg/kg) within 120 minutes of surgery start time.
  Interventions: Drug: Gentamicin, 5mg/kg; Drug: Ampicillin 2g; Drug: Gentamicin, 80 mg, 48hr
- 3b: +UCx No Oral options (7d) (Active Comparator): This group has a positive pre-operative urine culture with no oral antibiotic options based on culture sensitivities
  * 7 day course of an IV/Intramuscular (IM) antibiotic (proven effective on sensitivity profile)
  * Gentamicin (80 mg) preferred if sensitive
  * All patient receive ampicillin IV (2 g) and gentamicin IV (5 mg/kg) within 120 minutes of surgery start time.
  Interventions: Drug: Gentamicin, 5mg/kg; Drug: Ampicillin 2g; Drug: Gentamicin, 80 mg, 7d

INTERVENTIONS:
Drug: Nitrofurantoin 100 MG, 7d — 7 day course, 100 mg twice daily, PO
  Other Names: Macrobid
  Arms: 1b: Indwelling drains (7d); 2b: +UCx with Oral Options (7d)
Drug: Gentamicin, 5mg/kg — Peri-operative dose: 5 mg/kg of ideal body weight, IV
  Other Names: Gentamicin
Drug: Ampicillin 2g — Peri-operative dose: 2 grams, IV
Drug: Nitrofurantoin 100 mg, 48 hrs — 48 hour course, 100 mg twice daily, PO
  Other Names: Macrobid
  Arms: 1a: Indwelling drains (48 hr); 2a: +UCx with Oral Options (48hr)
Drug: Gentamicin, 80 mg, 7d — 7 day course, 80 mg daily, IM or IV
  Arms: 3b: +UCx No Oral options (7d)
Drug: Gentamicin, 80 mg, 48hr — 48 hour course, 80 mg daily, IM or IV
  Arms: 3a: +UCx No Oral options (48hr)

SUMMARY:
This study will be a multi-institutional randomized clinical trial of a short course of pre-operative antibiotic prophylaxis in addition to perioperative antibiotics prior to undergoing percutaneous nephrolithotomy. The select patient population will be those patients deemed to be at a moderately increased risk of postoperative infectious complications. These higher risk patients are those with indwelling urinary drainage tubes and those with a positive preoperative urine culture.

DETAILED DESCRIPTION:
This study will be a multi-institutional randomized clinical trial of a short course of pre-operative antibiotic prophylaxis in addition to perioperative antibiotics. Once patients have been identified and enrolled into the study, they will be grouped based on the sensitivity profiles of their positive urine culture or the presence of indwelling kidney drain tube (nephrostomy tube, nephroureteral stent, ureteral stent). Each of these groups will be individually randomized as follows:

Group 1) Kidney stone subjects with indwelling drain tube (nephrostomy tube or ureteral stent) and negative urine culture

Randomization:

* 7 day course of oral Macrobid (Nitrofurantoin) 100 mg twice daily + <24 hours perioperative intravenous (IV) antibiotics
* 48 hours perioperative oral Macrobid (Nitrofurantoin) 100mg twice daily + <24 hours perioperative IV antibiotics

Group 2) Kidney stone subjects with positive urine culture sensitive to oral antibiotics

Randomization:

* 7 day course of an oral antibiotic (proven effective on sensitivity profile) + <24 hours perioperative IV antibiotics
* 48 hours of an oral antibiotic (proven effective on sensitivity profile) + <24 hours perioperative IV antibiotics

Macrobid is preferred oral agent if shown to be effective per culture sensitivities. If patient has previous allergies to Macrobid and/or sensitivity profile indicates ineffectiveness of Macrobid, the one antibiotic will be provided in the order of choice: nitrofurantoin > sulfamethoxazole-trimethoprim > doxycycline> ciprofloxacin > keflex > cefpodoxime.

Group 3) Kidney stone subject with positive urine culture sensitive to only intravenous/intramuscular antibiotics (resistant to oral agents)

Randomization:

* 7 day course of an IV/Intramuscular (IM) antibiotic (proven effective on sensitivity profile) + <24 hours perioperative IV antibiotics
* 48 hours of an IV/IM antibiotic (proven effective on sensitivity profile) + <24 hours perioperative IV antibiotics peripherally inserted central catheter (PICC) line, IV or intramuscular injection for administration of antibiotics.

The participating institutions are academic medical centers in the United States and Canada that are part of the EDGE (Endourologic Disease Group of Excellence) research consortium, a research collaborative that has the goal of producing high quality, multi-institutional studies of nephrolithiasis. Separate IRB approvals will be obtained from each institution. University of California San Diego (UCSD) will be the coordinating institution. Member institution of EDGE maintain frequent email contact with one another and hold a monthly teleconference to discuss safety updates, interim results, issues with accrual, and modifications to research protocols and consents (if necessary).

Treatment Assignments:

Patients will be assigned based on a predetermined allocation sequence that will be generated by a computerized random number generator. Patients will be stratified by institution in permuted blocks of varying size. Only study staff at the coordinating institution (UCSD) will have access to the full allocation sequence. i.e. no clinical staff involved in recruiting and consenting patients for the study at UCSD or other participating institutions will have knowledge of the allocation sequence at their institution prior to enrollment of each patient. To further aid allocation concealment, the block size will be varied.

Standard of care procedures:

Patients will be identified based on clinic visits or hospital admission. All patients will be counseled on standard treatment options-extracorporeal shock wave lithotripsy (ESWL), percutaneous nephrolithotomy (PCNL) and ureteroscopy (URS). The discussion regarding treatment options and subsequent care will not deviate from routine care. Patients consenting for percutaneous nephrolithotomy (PCNL) will be considered for enrollment into the study and will be enrolled to have data collected prospectively. Patients will be consented prior to prescription of antibiotics and to the surgery for collection of demographic, disease, perioperative, and postoperative data. Abdominal pelvic computed tomography (CT), if not already obtained, will be used to delineate pre-operative stone size and for preoperative planning. If the patient does not consent to the study, the use of antibiotics will be based on routine clinical practice of the treating urologist. Both prophylaxis with preoperative antibiotics and no prophylaxis (i.e. periprocedural only) are considered standard of care.

Investigational portion of treatment:

Group 1 patients will be randomized to nitrofurantoin monohydrate/macrocrystalline 100 mg twice daily for 7 days prior to PCNL with the final day of prophylactic course being 1 day prior to surgery or to nitrofurantoin monohydrate/macrocrystalline 100mg twice daily for 48 hours prior to PCNL. Nitrofurantoin monohydrate/macrocrystalline is currently indicated for the treatment of acute uncomplicated urinary tract infections. Both groups will receive antibiotics the day of surgery-i.e. a dose of ampicillin intravenous (IV) (2 g) and gentamicin intravenous (IV) (5 mg/kg) within 120 minutes of surgery start time. Patients with penicillin allergy will receive vancomycin intravenous (IV) (1 g) instead of ampicillin and patients with gentamicin/aminoglycoside allergy will receive ceftriaxone intravenous (IV) (2 g) instead of gentamicin. Postoperative antibiotics in the absence of sepsis (see definition of sepsis below) will be <24 hours of IV antibiotics.

Group 2 patients will be randomized to either 7 days or 48 hours of oral antibiotics prior to the PCNL with the final day of prophylactic course being 1 day prior to surgery. Antibiotic choice will be determined by the culture sensitivity profile, with nitrofurantoin monohydrate/macrocrystalline 100 mg twice daily being the preferred agent if shown to be effective against the uropathogen(s). If patient has previous allergies to Macrobid and/or sensitivity profile indicates ineffectiveness of Macrobid, then one antibiotic will be provided in the following order: nitrofurantoin > sulfamethoxazole-trimethoprim > doxycycline> ciprofloxacin > keflex > cefpodoxime.

Antibiotics the day of surgery will be a dose of ampicillin IV (2g) and gentamicin IV (5mg/kg) within 120 minutes of surgery start time. Patients with penicillin allergy will receive vancomycin IV (1g) instead of ampicillin and patients with gentamicin/aminoglycoside allergy will receive ceftriaxone IV (2g) instead of gentamicin. Postoperative antibiotics in the absence of sepsis (see definition of sepsis below) will be <24 hours of IV antibiotics.

Group 3 patients will be randomized to either 7 days or 48 hours of an injectable (IV/IM) antibiotic prior to the PCNL with the final day of prophylaxis being 1 day before surgery. Antibiotic choice will be determined by the culture sensitivity profile.

Antibiotics the day of surgery will be a dose of same IV/IM antibiotic within 120 minutes of surgery start time. Postoperative antibiotics in the absence of sepsis (see definition of sepsis below) will be <24 hours of IV antibiotics.

Central randomization will take place with UCSD as the lead site. Randomization will occur in block randomization in block sizes of 10.

Standard of care procedures:

Patients will have PCNL performed in typical fashion, without deviation from standard of care. Per the usual practice of the treating surgeon, percutaneous access to the kidney will be obtained either by Interventional Radiology or by the operating surgeon. At the time of surgery, urine from the renal pelvis, urine from the bladder, and the stone itself will be sent for culture. Placement of renal drainage devices (ureteral stents, nephrostomy tubes, nephroureteral stents) will be left up to the discretion of the surgeon. Post-operatively, the patients will be admitted to the hospital and monitored per usual clinical procedure. Unless clinically indicated as described above, <24 hours of post-operative antibiotics will be prescribed. Labs will be obtained pre-operatively and on post-operative day 1 if the patient is admitted, and will include: complete blood count (CBC), basic metabolic panel (chem 7). Further laboratory tests will be dictated by the patients' clinical status as per the standard of care-i.e. for patients that exhibit signs of sepsis such as tachycardia (>90/min), low systolic blood pressure (<90 mmHg), fever > 38.3 Celsius, hypothermia <36 Celsius, altered mental status, respiratory rate >20 min or leukocytosis >12000 or leukopenia <4000, further urine culture, blood culture and serum lactate will be obtained.

The patient will be discharged from the hospital per the usual clinical protocols. Post-discharge the patient will be seen in clinic 1-12 weeks after surgery. Patients will undergo a non-contrast CT abdomen/pelvis, an abdominal plain radiograph, and/or a renal ultrasound during this postoperative period.

Demographic fields will be obtained preoperatively and include age, race, gender, American Society of Anesthesiologists (ASA) score (for comorbidity assessment), body mass index (BMI), and prior stone disease. Disease fields that will be obtained include stone size (maximal axial and coronal dimensions), degree of hydronephrosis (mild/moderate/severe), history of diabetes mellitus, history of cardiac disease, hypertension, prior urinary tract infection, history of bowel diversion, or neurogenic bladder.

Perioperative fields include OR (surgical) time, type of anesthesia, number of access tracts, use of internalized ureteral stent, nephrostomy tube, or nephroureteral stent, estimated blood loss, and intraoperative complications. Postoperative fields will include postoperative maximum body temperature, heart rate, respiratory rate, urine culture results, stone culture results, stone composition, white blood cell count, serum lactate, postoperative serum creatinine, need for admission to intensive care unit, hospital length of stay (LOS), and stone-free status at 1-12 week postoperative imaging. Patients will be followed during routine clinical visits as part of their continuing care.

ELIGIBILITY:
Age: >17 years of age

Gender: both men and women included. We anticipated enrolling a study population of approximately 60% men and 40% women based on a higher incidence of kidney stones among men in NHANES data.

Ethnic background: all ethnicities will be included in the study population and the specific ethnic diversity present in the study population will reflect the geographic distributions of the participating institutions.

Health status: see below for specific inclusion/exclusion criteria.

Inclusion criteria:

* Renal stone of any size for which PCNL is recommended
* Positive preoperative urine culture within 3 months
* Current internalized ureteral stent, nephrostomy tube, nephroureteral stent

Exclusion criteria

* Patients age <18
* Active pregnancy
* Patients receiving antibiotic doses (other than prescribed for the study) within the seven days preceding surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
postoperative sepsis | 30 days
  Sepsis will be defined by the 2012 International Guidelines for the Management of Severe Sepsis and Septic Shock where 2 or more of the following variables are present and temporally associated
  * Temp > 38.3C or <36C
  * Heart Rate > 90/min (at least 12 hrs after surgery)
  * Respiratory Rate >20/min (at least 12 hrs after surgery)
  * Altered mental status: defined as lack of orientation to either name, place or time/date
  * Systolic Blood Pressure (SBP) <90 mmHg, Mean Arterial Pressure <70 mmHg, or SBP decrease >40 mmHg in adults
  * White blood cell (WBC) > 12000 or <4000

SECONDARY OUTCOMES:
rate of nonseptic bacteruria | 30 days
  -non septic bacteria is the presence of any colony forming units on urine culture where sepsis is not present
stone-free rate | 30 days
  stone free defined as absence of kidney stone on all post-operative imaging (plain kidney-ureter-bladder X-ray or renal ultrasound or computed tomography)
Length of hospital stay | 30 days
  hospital day defined as any inpatient stay < or = 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
RedCap Password Protected Data Share System

REFERENCES:
- [Result] de la Rosette J, Assimos D, Desai M, Gutierrez J, Lingeman J, Scarpa R, Tefekli A; CROES PCNL Study Group. The Clinical Research Office of the Endourological Society Percutaneous Nephrolithotomy Global Study: indications, complications, and outcomes in 5803 patients. J Endourol. 2011 Jan;25(1):11-7. doi: 10.1089/end.2010.0424. PMID 21247286
- [Result] Korets R, Graversen JA, Kates M, Mues AC, Gupta M. Post-percutaneous nephrolithotomy systemic inflammatory response: a prospective analysis of preoperative urine, renal pelvic urine and stone cultures. J Urol. 2011 Nov;186(5):1899-903. doi: 10.1016/j.juro.2011.06.064. Epub 2011 Sep 23. PMID 21944106
- [Result] Kumar S, Bag S, Ganesamoni R, Mandal AK, Taneja N, Singh SK. Risk factors for urosepsis following percutaneous nephrolithotomy: role of 1 week of nitrofurantoin in reducing the risk of urosepsis. Urol Res. 2012 Feb;40(1):79-86. doi: 10.1007/s00240-011-0386-6. Epub 2011 May 13. PMID 21567157
- [Result] Bag S, Kumar S, Taneja N, Sharma V, Mandal AK, Singh SK. One week of nitrofurantoin before percutaneous nephrolithotomy significantly reduces upper tract infection and urosepsis: a prospective controlled study. Urology. 2011 Jan;77(1):45-9. doi: 10.1016/j.urology.2010.03.025. Epub 2010 Jun 8. PMID 20570319
- [Result] Wolf JS Jr, Bennett CJ, Dmochowski RR, Hollenbeck BK, Pearle MS, Schaeffer AJ; Urologic Surgery Antimicrobial Prophylaxis Best Practice Policy Panel. Best practice policy statement on urologic surgery antimicrobial prophylaxis. J Urol. 2008 Apr;179(4):1379-90. doi: 10.1016/j.juro.2008.01.068. Epub 2008 Feb 20. PMID 18280509
- [Derived] Sur RL, Krambeck AE, Large T, Bechis SK, Friedlander DF, Monga M, Hsi RS, Miller NL, Chew BH, Lange D, Knudsen B, Sourial MW, Humphreys MR, Stern KL, Shah O, Abbott JE, Abedi G. A Randomized Controlled Trial of Preoperative Prophylactic Antibiotics for Percutaneous Nephrolithotomy in Moderate to High Infectious Risk Population: A Report from the EDGE Consortium. J Urol. 2021 May;205(5):1379-1386. doi: 10.1097/JU.0000000000001582. Epub 2020 Dec 28. PMID 33369488